CLINICAL TRIAL: NCT06010615
Title: Relative Dose Intensity of Adjuvant Chemotherapy in Older Women With ER+ HER2- Breast Cancer.
Acronym: BREASTOLD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/785
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Localized breast cancers are defined as high-risk when they include lymph node involvement, Ki67 >30%, vascular emboli, low hormone receptor expression, or an unfavorable genomic signature result.

Under these conditions, sequential adjuvant chemotherapy with taxanes and anthracyclines is recommended.

Patients over 75 years of age receiving adjuvant chemotherapy are at greater risk of side-effects, which may necessitate dose reductions and a reduction in the intensity of chemotherapy. For curative adjuvant treatment, it is recommended to maintain a relative dose intensity (RDI) > 85%. A few publications have demonstrated the prognostic impact of a relative dose intensity < 85% for patients aged over 65. For several years now, the need for a specific assessment of elderly patients has been emphasized, prior to initiating oncological treatment (G8 score, onco-geriatric consultation).

This study is a retrospective descriptive study of patients aged over 75 treated with adjuvant chemotherapy from 01/01/2012 to 01/01/2020 for RH+ HER2 - breast cancer in Franche Comté.

Thus the investigators wish to identify patients at risk of receiving sub-optimal relative dose intensity, in order to guide early and targeted supportive care or geriatric co-management interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 75 or over
* Patient with localized RH+HER2- breast cancer
* Patient treated with adjuvant chemotherapy in Franche Comté between January 2012 and December 2019

Exclusion Criteria:

* Age < 75
* Patient with metastatic breast cancer
* Patient who received neoadjuvant chemotherapy
* HER2+ breast cancer patient
* Breast cancer patient with missing or negative hormonal status
* Patient with localized recurrence of breast cancer with indication for new adjuvant therapy

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 75 and over with RH+ HER2- breast cancer who received adjuvant chemotherapy between 01/01/2012 and 01/01/2020, within the Regional Cancer Network of Bourgogne-Franche-Comté - oncoBFC
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving relative dose intensity (RDI) <85% | 01/01/2012 to 31/12/2019

IPD SHARING:
Plan to Share IPD: No